CLINICAL TRIAL: NCT06796348
Title: Multi-center, 1:1 Randomized, Stratified, Parallel-group, Non-inferiority Clinical Trial of Small Thyroid Cancers Treated with Hemithyroidectomy or Radiofrequency Ablation.
Brief Title: Radiofrequency Ablation Versus Hemithyroidectomy of Small Thyroid Cancers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFARCT8200
Record Dates: First submitted 2024-12-17; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer
Keywords: Radiofrequency ablation; Hemithyroidectomy; thyroid cancer; Differentiated thyroid carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Radiofrequency Ablation; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery of thyroid cancer (Active Comparator)
  Interventions: Procedure: Surgery
- RFA of thyroid cancer (Experimental)
  Interventions: Procedure: Radiofrequency ablation alone

INTERVENTIONS:
Procedure: Radiofrequency ablation alone — RFA of a cancer in the thyroid gland.
  Arms: RFA of thyroid cancer
Procedure: Surgery — Hemithyroidectomy of the thyroid lobe with cancer
  Arms: Surgery of thyroid cancer

SUMMARY:
This is a multicenter randomized controlled trial including patients with small (<2 cm) suspected or confirmed thyroid cancers. Patients are included after informed consent and randomized to one of two treatments. One treatment is a standard henithyroidectomy and the second treatment is radiofrequency ablation (RFA) of the specific tumor. The investigators will evaluate initial outcome of the allocated treatment, thyroid hormonal function, oncologic safety, quality of life, and treatment costs in a follow-up period of five years after treatment.

The overall aim of the study is to improve patient's health by reducing the number of operations on small thyroid cancers. In patients with these small tumors, the long-term adverse outcome may be higher than possible benefits from the operation. For participants undergoing surgical treatment with HT, the investigators will measure final histology and both beneficial and adverse outcome from the operation. For participants undergoing RFA, the investigators expect to reduce the need for thyroid hormonal substitutions, reduce the surgical adverse outcomes, reduce treatment costs and increase QoL without a reduction in oncologic safety and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Single tumor in the thyroid gland with a FNAB suspecious of cancer or diagnostic of cancer (category V or VI in the Bethesda system)
* tumor size of less than 2 cm in all dimensions.

Exclusion Criteria:

* suspicion of disseminated disease because of PET-positive lymph nodes ; suspect lymph-nodes by ultrasonography (US); or signs of capsular invasion of the tumor OR
* tumor not eligible for RFA treatment because of high-risk location; previous thyroid surgery; concomitant hyperparathyroidism (ionized calcium > 1.32 mmol/L and PTH > 6 pmol//L ) OR
* if the patient is pregnant OR
* If the patient is unable to give informed consent.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Uncomplicated initial treatment (yes/no) | One month after randomization.
  Uncomplicated treatment is defined as a composite endpoint (dichotomous; yes/no) with none of the following adverse outcomes within the first month after treatment/surgery:
  1. short or long-term affection of the recurrent laryngeal nerve (RLN) based on laryngoscopy,
  2. infection with a need for surgical treatment,
  3. capsule rupture or bleeding with a need for operation,
  4. prolonged hospital stay (more than one night),
  5. any other reason for a secondary surgical intervention on the neck.

SECONDARY OUTCOMES:
Oncologic | 5 years after randomization.
  Any oncologic events with either recurrence of disease in the thyroid gland or lymph node metastasis are included (dichotomous; yes/no). Developing disease in the contralateral side of the thyroid gland will also be described and evaluated and possibly treated. However, contralateral disease will not be classified as adverse outcome after initial treatment but rather classified as new disease (dichotomous; yes/no).
Endocrinological 1 | At three months, 1, 2, 3, 4 and 5 years after randomization.
  The need for substitutional treatment with thyroid hormones (dichotomous; yes/no) is included as secondary endpoint.
Patient-reported outcome 1 | At randomization (baseline), and at three months, 1, 2, 3, 4, and 5 years after randomization.
  A patient reported outcome is collected with use of the thyroid specific questionnaire ThyPRO-39 (continuous outcome).
Health economics | At 5 years after randomization.
  Collective costs for treatment with a HT operation in general anesthesia and an in-hospital stay is much more expensive than RFA treatment in the outpatient clinic. The relation between total costs for HT versus RFA are close to 5:1 and all treatment related costs will be collected during the trial.
Patient-reported outcome 2 | At randomization (baseline), and at three months, 1, 2, 3, 4, and 5 years after randomization.
  A patient reported outcome is collected with use of the thyroid specific questionnaire Voice Related QoL (V-RQoL) (continuous outcome).

OTHER OUTCOMES:
Endocrinological 2 | At randomization (baseline), and at three months, 1, 2, 3, 4 and 5 years after randomization.
  Thyroid hormones are evaluated by biochemical measurements (mU/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data of the results from the primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting information and IPD will be available by January 2026 and until January 2030.
Access Criteria: By contact to the primary investigator and trial manager.